CLINICAL TRIAL: NCT02404337
Title: Betaine METABOLISM OF PATIENTS With Homocystinuria
Acronym: HCTBETAINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P130908
Record Dates: First submitted 2015-03-06; First posted 2015-03-31 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2018-02

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria | interventions — Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 mg/kg of Betaine (Experimental): Dose 1 : 100 mg/kg of Betaine
  Interventions: Drug: Betaine
- 250 mg/kg of Betaine (Experimental): Dose 2 : 250 mg/kg of Betaine
  Interventions: Drug: Betaine

INTERVENTIONS:
Drug: Betaine

SUMMARY:
Oral treatment with betaine is conventionally used for patients with inherited homocystinurias.

These conditions include a first group of patients with a cystathionine β-synthase (CBS) deficiency and a second group of patients with remethylation defects.

The aim of betaine therapy is to reduce level of total plasma homocysteine. Daily dosages and rhythm of administration proposed in the literature vary between 100 to 250 mg / kg / d in 2 to 4 doses. These dosages are not based on validated data and several publications mention much higher dosages particularly when total homocysteine is not controlled. These practices may be unnecessary or even detrimental given the fact that high doses of betaine could for example lead to secondary folate deficiency.

DETAILED DESCRIPTION:
Oral treatment with betaine is conventionally used for patients with inherited homocystinurias.

These conditions include a first group of patients with a cystathionine β-synthase (CBS) deficiency and a second group of patients with remethylation defects.

The aim of betaine therapy is to reduce level of total plasma homocysteine. Daily dosages and rhythm of administration proposed in the literature vary between 100 to 250 mg / kg / d in 2 to 4 doses. These dosages are not based on validated data and several publications mention much higher dosages particularly when total homocysteine is not controlled. These practices may be unnecessary or even detrimental given the fact that high doses of betaine could for example lead to secondary folate deficiency.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 year and children <18 years,
* homocystinuria confirmed enzymatically or molecularly divided into 2 groups:

  * CBS deficiency remethylation defects (CbIC defect and MTHFR deficiency)
* Diagnosis of homocystinuria since more than 1 year
* Continuous treatment of hyperhomocysteinemia in the last 12 months

Exclusion Criteria:

* Deficits in cystathionine beta-synthase B6-responsive
* pregnancy
* breast-feeding
* Young pubescent girls not using effective contraception

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Plasma level of total homocysteine upon oral treatment with Betaine at 100 mg / kg / day compared with 250 mg / kg / day in the same individual. | 10 weeks - at the end of follow-up of each patient
  The assay technique used is MS/MS validated according to ISO standard 1589. Samples will be frozen and analysed at the end of follow-up of the study. Freezing does not affect the validity of the technique used.

SECONDARY OUTCOMES:
Measurement of dimethylglycine plasma level following the loading dose of 100 mg / kg of betaine compared in the same person with the dose of 250 mg / kg. | 10 weeks - at the end of follow-up of each patient
Measurement of sarcosine plasma level following the loading dose of 100 mg / kg of betaine compared in the same person with the dose of 250 mg / kg. | 10 weeks - at the end of follow-up of each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France

REFERENCES:
- [Result] Imbard A, Toumazi A, Magreault S, Garcia-Segarra N, Schlemmer D, Kaguelidou F, Perronneau I, Haignere J, de Baulny HO, Kuster A, Feillet F, Alberti C, Guilmin-Crepon S, Benoist JF, Schiff M. Efficacy and pharmacokinetics of betaine in CBS and cblC deficiencies: a cross-over randomized controlled trial. Orphanet J Rare Dis. 2022 Nov 14;17(1):417. doi: 10.1186/s13023-022-02567-4. PMID 36376887